CLINICAL TRIAL: NCT04475432
Title: Randomized, Controlled, Multicenter, Double-Masked, Parallel, Phase 2b/3 Trial to Evaluate the Safety and Efficacy of TP-03 for the Treatment of Demodex Blepharitis
Brief Title: Safety and Efficacy of TP-03 for the Treatment of Demodex Blepharitis
Acronym: Saturn-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS-009
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Blepharitis
Keywords: Demodex
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Intervention Model Description: Active arm: TP-03 0.25%
  Control arm: Vehicle of TP-03
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment assignment will be unknown to the study participant, investigators and site staff performing study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): TP-03, lotilaner ophthalmic solution, 0.25%, administered topically twice a day for approximately 43 days
  Interventions: Drug: TP-03, 0.25%
- Control (Placebo Comparator): Vehicle of TP-03 ophthalmic solution, administered topically twice a day for approximately 43 days
  Interventions: Drug: TP-03 Vehicle

INTERVENTIONS:
Drug: TP-03, 0.25% — TP-03, lotilaner ophthalmic solution, 0.25%, administered twice a day
  Other Names: Lotilaner ophthalmic solution, 0.25%
  Arms: Active
Drug: TP-03 Vehicle — Vehicle of TP-03 ophthalmic solution, administered twice a day
  Arms: Control

SUMMARY:
The purpose of this study is to compare the safety and efficacy of TP-03, 0.25%, an eyedrop, to its vehicle control for the treatment of blepharitis due to Demodex, a microscopic mite frequently found in human hair follicles. The hypothesis for the study is the proportion of participants cured at Day 43 with treatment by TP-03, 0.25%, is greater than the proportion cured by treatment with its vehicle.

DETAILED DESCRIPTION:
This Phase 2b/3 study is a randomized, controlled, multicenter, double-masked, parallel trial to compare the safety and efficacy of TP-03, 0.25%, to vehicle control for the treatment of Demodex blepharitis. The primary objective of the study is to assess the safety and efficacy of TP-03 compared to its vehicle from Day 1 to Day 43 in adult participants with mild to severe Demodex blepharitis. The primary efficacy endpoint will be cure based upon collarettes. Safety will be determined by assessing adverse effects related to the treatment as well as evaluating any changes in visual acuity, intraocular pressure, slit lamp biomicroscopy and dilated ophthalmoscopy findings.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol
* Meet all of the following criteria in at least one eye: Have more than 10 lashes with collarettes present on the upper lid; have at least mild erythema of the upper eyelid margin; have an average Demodex density, upper and lower eyelids combined, of 1.5 or more mites per lash

Exclusion Criteria:

* Have used lid hygiene products within 14 days of Screening or unwilling to forego the use of lid hygiene products during the study
* Have worn contact lenses within 7 days of Screening or be unwilling to forego contact lens wear during the study
* Have used artificial eyelashes or eyelash extensions within 7 days of Screening or be unwilling to forego their use during the study
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wirta, MD, Principal Investigator — Eye Research Foundation
Locations (15):
- United States (15):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Visionary Eye Institute, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Washburn Research LLC, Indianapolis, Indiana
  - The Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Ophthalmology Associates, St Louis, Missouri
  - Oculus Research, Inc at EyecareCenter, Raleigh, North Carolina
  - Vita Eye Clinic, Shelby, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Total Eye Care, P.A., Memphis, Tennessee
  - Alpine Research Organization, Layton, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeu E, Wirta DL, Karpecki P, Baba SN, Holdbrook M; Saturn I Study Group. Lotilaner Ophthalmic Solution, 0.25%, for the Treatment of Demodex Blepharitis: Results of a Prospective, Randomized, Vehicle-Controlled, Double-Masked, Pivotal Trial (Saturn-1). Cornea. 2023 Apr 1;42(4):435-443. doi: 10.1097/ICO.0000000000003097. Epub 2022 Aug 10. PMID 35965392

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: TP-03, lotilaner ophthalmic solution, 0.25%, administered twice a day
- Control: Vehicle of TP-03 topical ophthalmic solution, administered twice a day
Period: Overall Study
Arm/Group | Active | Control
Started | 212 | 209
Completed | 208 | 203
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 212 | 209 | 421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 65 | 151
  >=65 years | 126 | 144 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (12.09) | 67.8 (12.63) | 67.0 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 117 | 240
  Male | 89 | 92 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 198 | 198 | 396
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 16 | 27
  White | 195 | 187 | 382
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 212 | 209 | 421

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Cured Based on a Collarette Score at Day 43.
Description: The proportion of participants cured where cure is defined as 0-2 lashes with collarettes on the upper eyelid of the analysis eye.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values.
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion cured
Arm/Group | Active | Control
Number analyzed (Participants) | 212 | 209
Proportion cured | 0.439 (0.034) | 0.072 (0.018)

2. Secondary Outcome: The Proportion of Participants With Eradication of Demodex Mites in the Analysis Eye at Day 43
Description: The proportion of participants with Demodex mites eradicated at Day 43 where eradication is defined as a mite density of 0 mites/lash for the analysis eye. The mite density is obtained by epilating four of more lashes and dividing the number of mites observed under the microscope by the number of lashes.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion eradicated
Groups:
- Active: TP-03, lotilaner ophthalmic solution, 0.25%, administered topically twice a day
- Control: Vehicle of TP-03 ophthalmic solution, administered topically twice a day
Arm/Group | Active | Control
Number analyzed (Participants) | 212 | 209
Proportion eradicated | 0.677 (0.032) | 0.173 (0.026)

3. Secondary Outcome: Proportion of Participants Cured Based on a Composite Collarette and Erythema Score of 0 in the Analysis Eye at Day 43.
Description: The proportion of participants cured where cure is defined as a composite of the collarettes, 0-2 lashes with collarettes on the upper eyelid of the analysis eye, and normal lid margin erythema for the upper eyelid of the analysis eye at Day 43.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values.
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion cured
Arm/Group | Active | Control
Number analyzed (Participants) | 212 | 209
Proportion cured | 0.139 (0.024) | 0.01 (0.007)

ADVERSE EVENTS:
Time Frame: 57 days
Description: Corresponds to the standard definition.
Groups:
- Active: TP-03, lotilaner ophthalmic solution, 0.25%, administered twice a day for approximately 43 days
- Control: Vehicle of TP-03 topical ophthalmic solution, administered twice a day for approximately 43 days
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/209
Serious Adverse Events (participants affected / at risk) | 3/212 | 1/209
Other Adverse Events (participants affected / at risk) | 37/212 | 39/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=212) | Control (N=209)
COVID-19 (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=212) | Control (N=209)
Visual acuity reduced (Eye disorders) | 6 | 6
Eye pain (Eye disorders) | 3 | 3
Eye discharge (Eye disorders) | 3 | 2
Chalazion (Eye disorders) | 1 | 3
Vision blurred (Eye disorders) | 2 | 2
Eye pruritus (Eye disorders) | 1 | 2
Swelling of eyelid (Eye disorders) | 1 | 2
Instillation site pain (General disorders) | 25 | 16
Instillation site pruritus (General disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is specified in the protocol that the data generated in this clinical trial, all related information and any materials containing such data and information are the exclusive property of Tarsus Pharmaceuticals, Inc. and are confidential to Tarsus Pharmaceuticals. Also, the investigator or other study-related personnel may not disclose to anyone or use any data, information or materials related to this clinical trial without the express written consent of Tarsus Pharmaceuticals.

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04475432/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04475432/SAP_003.pdf